CLINICAL TRIAL: NCT05958901
Title: A Observational Study in Chinese Patients With Pulmonary Hypertension (PH)
Brief Title: Pulmonary Hypertension Observational Study
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, zili zhang, Zili Zhang, The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: Pulmonary Hypertension of GIRH
Record Dates: First submitted 2023-07-12; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pulmonary hypertension
  Interventions: Other: pulmonary hypertension
- healthy

INTERVENTIONS:
Other: pulmonary hypertension — The final outcome observed was a diagnosis of pulmonary hypertension.
  Groups: pulmonary hypertension

SUMMARY:
The purpose of this study is to establish the large PH cohort and biological database in China, aiming for precision medicine to optimize diagnosis and treatment choices.

ELIGIBILITY:
Inclusion Criteria:

* PH group: When the mean pulmonary artery pressure is greater than 25mmHg at rest or greater than 30mmHg during exercise.
* Signed informed consent obtained prior to participations with the ability to comply with protocol and be available for study visits over 5 years.

Exclusion Criteria:

* Acute exacerbation in the past 3 months Having other respiratory diseases with massive lung tissue destruction such as severe bronchiectasis and tuberculosis, etc.
* Serious uncontrolled diseases thoracic or abdominal surgery in the last 3 months.
* Eye surgery in the last three months.
* Retinal detachment myocardial infarction in the last 3 months.
* Admission to hospital for any cardiac condition in the last month.
* Heart rate over 120 beats per minute.
* Antibacterial chemotherapy for tuberculosis pregnant or breast feeding.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a observational prospective longitudinal cohort study to to establish the large PH cohort and biological database in China, including PH subjects( n= 5000) and healthy subjects (n= 5000). Sites Investigators will be respiratory physicians working in the respiratory department of our sites, which must be tier 2 or tier 3 hospitals in China, with the equipment and ability to conduct right heart catheterization(RHC). Patients must meet all the inclusion criteria and none of the exclusion criteria. No additional investigational drugs will be applied to the patients. Statistical analysis will be conducted by epidemiology & statistics work group from Chinese Academy of Sciences, using SAS and R software. Paper-based questionnaire administration will also be used. Questionnaire variables will be checked before data entry. During the study, PI will be in charge of the monitoring of the whole procedure.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
mean pulmonary arterial pressure | 12 months
  For an adult at sea level, when the mean pulmonary arterial pressure is greater than 25 mmHg at rest or greater than 30mmHg during exercise.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes